CLINICAL TRIAL: NCT02911688
Title: Effect of Gamma Tocopherol Enriched Supplementation on Response to Inhaled O3 Exposure
Acronym: Gammoz
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-1938; 4R01ES023349-04 (NIH)
Record Dates: First submitted 2016-09-08; First posted 2016-09-22 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-02

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — gamma-Tocopherol; Vitamin E; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Safflower oil, taken in 2 capsules every 12 hours for a total of 4 doses
  Interventions: Drug: Placebo
- gamma tocopherol (Active Comparator): gamma tocopherol 1400 mg, taken as 2 700 mg capsules every 12 hours for a total of 4 doses
  Interventions: Drug: gamma tocopherol

INTERVENTIONS:
Drug: gamma tocopherol — The effect of supplemental with gamma tocopherol on O3 response will be assessed using the difference pre and after γT dosing.
  Other Names: Vitamin E
  Arms: gamma tocopherol
Drug: Placebo — The effect of supplemental with gamma tocopherol on O3 response will be assessed using the difference pre and after placebo dosing.
  Other Names: Safflower oil
  Arms: placebo

SUMMARY:
To study the effects of 1200mg gamma tocopherol, a form of vitamin E, given daily on the response of the airway in mild asthmatics after exposure to ozone (O3)

DETAILED DESCRIPTION:
Allergic asthma (AA) is the most commonly encountered respiratory disease in children and adults in the United States and is a leading cause of morbidity worldwide. Among the most disruptive expressions of disease in AA is acute asthma exacerbation. The Center for Disease Control (CDC) lists ambient air pollutants and environmental tobacco smoke as among the most common triggers for acute asthma exacerbation. Ozone (O3) is the most commonly encountered ambient air pollutant in the US.

Increased oxidative stress and decreased antioxidant capability have been observed in asthmatics. These pollutants are pro-inflammatory and are associated with increased oxidative stress, which would exacerbate reactive oxygen and reactive nitrogen species (ROS and RNS)-induced injury in asthmatics. O3 injures epithelial cells, releasing secondary mediators which activate inflammatory cells, in part by ligation of Toll-like receptor 4 (TLR4), the primary receptor for lipopolysaccharide (LPS). TLR4 activation of inflammatory cells activates (nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB) and induces oxidative stress. O3 and LPS has been associated with exacerbation of asthma, and the investigators have reported that O3 and LPS augments allergic airway inflammation in allergic asthmatics (AA). Development of interventions to mitigate these responses will greatly decrease disease morbidity. Given the role that oxidants play in the pathophysiology of asthma exacerbation, defects in antioxidant levels would increase risk for acute asthma exacerbation. Nutritional deficiencies in vitamin E, ascorbate and selenium have been linked to asthma severity, and asthmatics have decreased antioxidant levels in airway fluid. It has been shown that vitamins C and E are decreased in airway fluids of asthmatics. Additionally, genetic factors may increase risk for oxidant induced exacerbation of asthma. Many investigators have reported that persons who are homozygous for the null polymorphism of the Glutathione-S-Transferase Mu1 (GSTM1) gene and unable to produce GSTM1 protein (the GSTM1 null genotype) have increased risk of acute pollutant-induced exacerbation of asthma. This lab has shown in healthy volunteers that the GSTM1 null genotype is associated with increased inflammatory response to O3, with no impact on the nociceptive response to this pollutant.

Other researchers have shown that the GSTM1 null genotype is associated with increased response to secondhand tobacco smoke, diesel exhaust, and other particulate matter components. Romieu et al demonstrated that children with asthma in Mexico City had increased susceptibility to O3-induced exacerbations if they had the GSTM1 null genotype. This group also found that GSTM1 null AAs selectively benefited from antioxidant intervention. The GSTM1 null genotype is found in 20-40% of the population, and may be overrepresented in allergic populations. Taken together, these observations show that the sizable GSTM1 null population is at risk for pollutant-induced airway disease, and that antioxidant intervention targeting the action of ROS and RNS will benefit asthmatics and especially GSTM1 null asthmatics.

A non-exclusive list of proposed antioxidants includes radical scavengers such as ascorbate, a-tocopherol (aT), y-tocopherol (γT) or inducers of Nuclear factor erythroid-2-related factor 2 (NRF2), which activate NRF2 with subsequent broad upregulation of acute phase II and antioxidant proteins. These agents are available in naturally occurring foods and as nutritional supplements. A number of animal, cell culture and epidemiological studies support the idea that antioxidant supplementation is useful in allergic airway disease. However, despite these studies and widespread public and scientific enthusiasm regarding use of such agents in asthmatics, there are scant human data to support or refute the use of such interventions for either acute or chronic allergic airways disease.

Gamma tocopherol has both radical scavenging and anti-inflammatory actions which may play important roles in decreasing pollutant-induced and allergic injury to the airway. Like other isoforms of vitamin E, γT is a potent ROS scavenger and is also a powerful nucleophile that traps electrophiles such as peroxynitrite in lipophilic compartments. One mechanism by which γT is cytoprotective is scavenging of RNS at the un-substituted C-5 position on the hydroxy-chroman ring of γT to form 5-NO-γ-tocopherol (5-NO-γT). Overall, vitamin E provides general protection of DNA, lipids and proteins from radical stress. An example of such protection is shown in rodent studies of prostate cancer in which intake of γT is associated with decreased DNA methylation of CpG rich regions of the NRF2. NRF2 is a master regulator of numerous cytoprotective antioxidant enzymes.

Supplementation with γT also prevents protein nitration and attenuates loss of plasma vitamin C in plasma in a rodent peritonitis model of inflammation. The investigators have also shown that γT inhibits Cyclooxygenase (COX)-2 and 5-Lipoxygenase (LO) in LPS-stimulated macrophages and interleukin (IL)-1b stimulated epithelial cells. These actions are mediated primarily by the γT metabolite 2, 7, 8-trimethyl-2S-(.-carboxyethyl)-6-hydroxychroman (γ-CEHC) which requires hydroxylation of the γ-methyl group of γT by cytochrome P450 (CYP450). In carrageenan- induced inflammation in male Wistar rats, γT decreases prostaglandin (PGE2) and leukotriene (LTB4) production, suggesting that LO-mediated production of leukotrienes may also be inhibited by γT. Tocopherols, including γT, also modulate gene expression of a number of inflammatory genes. Thus, γT and other tocopherols decrease production of a number of pro-inflammatory cytokines at the transcriptional level.

In animals, it has also been shown that gamma tocopherol reduces baseline eosinophilia in the airway. In early phase I studies of gamma tocopherol-enriched mixed tocopherols (γT-mT) the investigators have shown that γT-mT inhibits monocyte induced cytokine production, decreases baseline nitrosative stress, and inhibits LPS eosinophil and neutrophil influx in healthy volunteers.

SUMMARY:

There is widespread opinion that antioxidant nutrients like gamma tocopherol ( γT, a form of Vitamin E) are an untapped and inexpensive intervention for environmentally triggered acute asthma. However, there is a crucial gap in evidence-based support of such interventions in asthma. A lack of coordinated research assessing specific antioxidant regimens from preclinical, phase I and phase II studies impedes development of phase III antioxidant trials in asthmatic populations. It is also unclear which physiological endpoints are most relevant in such studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 of both genders
2. Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy
3. History of episodic wheezing, chest tightness, or shortness of breath consistent with asthma, or physician diagnosed asthma.
4. Positive methacholine test. A positive test is defined as a provocative concentration of methacholine of 10 mg/ml or less producing a 15% fall in forced expiratory volume in 1 second (FEV1) (PC20 methacholine) by the method used in a separate screening protocol or a pre and post bronchodilator challenge used to determine reversible lung function. Reversibility is confirmed with a 10-12% increase in FEV1 15 minutes after inhaling 4 puffs of albuterol with a spacer. Reversibility is used in the same separate screening protocol; or a clinical history of asthma after the age of 6.
5. FEV1 of at least 80% of predicted and FEV1/Forced Vital Capacity (FVC) ratio of at least .70 (without use of bronchodilating medications for 12 hours or long acting beta agonists for 24 hours), consistent with lung function of persons with no more than mild episodic or mild persistent asthma.
6. Allergic sensitization to at least one of the following allergen preparations: (House Dust Mite f, House dust mite p, Cockroach, Tree mix, Grass Mix, Weed Mix, Mold Mix 1, Mold Mix 2, Rat, Mouse, Guinea Pig, Rabbit, Cat or Dog) confirmed by positive immediate skin test response; or a clinical history consistent with seasonal or perennial allergy symptoms.
7. Symptom Score (this will be submitted as an attachment) no greater than 20 (out of a possible 60) for total symptom score with a value no greater than 3 for any one score. No more than one score may be greater or equal than 3.
8. subjects must be willing to avoid caffeine for 12 hours prior to all visits. Methacholine challenge and allergy skin testing are performed as part of IRB 98-0799, which a subject must complete in order to be considered for this protocol.
9. for subjects who are prescribed inhaled corticosteroids (ICS). These volunteers must be able to come off of the ICS for 2 weeks without increased symptoms or increased need for beta agonist rescue medication prior to screening and throughout the course of the study.

   -

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency, history of tuberculosis
2. Physician directed emergency treatment for an asthma exacerbation within the preceding 3 months
3. Moderate or Severe asthma
4. Exacerbation of asthma more than 2x/week which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
5. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
6. Viral upper respiratory tract infection within 4 weeks of challenge.
7. Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 4 weeks of challenge.
8. Severe asthma
9. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
10. Medications which may impact the results of the O3 exposure, interfere with any other medications potentially used in the study (to include systemic steroids, beta antagonists, non-steroidal anti-inflammatory agents)
11. Any history of smoking in the year prior to study enrollment; lifetime smoking history > 10 pack years
12. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma
13. Allergy/sensitivity to study drugs, or their formulations.
14. Known hypersensitivity to methacholine or to other parasympathomimetic agents
15. History of intubation for asthma
16. Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch, condoms).
17. Abnormal Prothrombin Time (PT) or activated Partial Thromboplastin Time (aPTT) values at screening or during the treatment period. Normal values will be those published by the clinical lab (Labcorp, INC).
18. Any bleeding disorder
19. Orthopedic conditions which would prevent the volunteer from performing moderate exercise on a treadmill.
20. Radiation exposure history will be collected. Subjects whose exposure history within the past twelve months would cause them to exceed their annual limits will be excluded.

    -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, Principal Investigator — UNC
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were screened for eligibility between September 2016 and November 2018 at the Center for Environmental Medicine, Asthma and Lung Biology at the University of North Carolina at Chapel Hill.
Pre-assignment Details: 18 volunteers were randomized
Groups:
- Placebo Then Gamma T: Participants first received safflower oil, taken in two 700 mg capsules every 12 hours for a total of 4 doses followed by a washout period of at least 3 weeks. Then they received gamma tocopherol-enriched supplement taken in two 700 mg capsules (total of 1200 mg of gamma tocopherol) every 12 hours for a total of 4 doses.
- Gamma Tocopherol Then Placebo: Participants first received gamma tocopherol-enriched supplement taken in two 700 mg capsules (total of 1200 mg of gamma tocopherol) every 12 hours for a total of 4 doses, followed by a washout period of at least 3 weeks. They then received safflower oil, taken in two 700 mg capsules every 12 hours for a total of 4 doses.
Period: First Intervention
Arm/Group | Placebo Then Gamma T | Gamma Tocopherol Then Placebo
Started | 9 | 9
Received Intervention | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout
Arm/Group | Placebo Then Gamma T | Gamma Tocopherol Then Placebo
Started | 9 | 9
Completed | 8 | 7
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Placebo Then Gamma T | Gamma Tocopherol Then Placebo
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Gamma T: Safflower oil, taken in 2 capsules every 12 hours for a total of 4 doses followed by a washout period of at least 3 weeks and then gamma tocopherol will be taken as 2 gel tabs (1200 mg/dose) every 12 hours for a total of 4 doses.
- Gamma Tocopherol Then Placebo: Gamma tocopherol will be taken 2 gel tabs (1200 mg/dose) every 12 hours for a total of 4 doses followed by a washout period of at least 3 weeks followed by safflower oil, taken in 2 capsules every 12 hours for a total of 4 doses.
- Total: Total of all reporting groups
Arm/Group | Placebo Then Gamma T | Gamma Tocopherol Then Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sputum Percent Neutrophils (%PMN) Following Ozone Exposure
Description: Participants provide induced sputum samples before and 6 hours after Ozone exposure for measurements of inflammatory cells. The analysis will determine if gamma tocopherol pre-treatment reduces ozone-induced sputum percent neutrophils compared to placebo pre-treatment.
Time Frame: baseline and 6 hours post-ozone exposure
Population: Due to variability in quality of induced sputum samples, paired assessments of pre and post-ozone sputum endpoints were limited to 7 volunteers.
Measure: Mean (Standard Deviation); unit: percent neutrophils
Groups:
- Gamma Tocopherol (N=7): gamma tocopherol 1400 mg, taken as two 700 mg capsules every 12 hours for a total of 4 doses
- Placebo (N=7): Safflower oil, taken in 2 capsules every 12 hours for a total of 4 doses
Arm/Group | Gamma Tocopherol (N=7) | Placebo (N=7)
Number analyzed (Participants) | 7 | 7
percent neutrophils | 34.1 (20.2) | 36.5 (20.2)

2. Secondary Outcome: Change in Sputum Percent Eosinophils From Baseline Following Ozone Exposure
Description: The investigators assessed induced sputum cellularity at baseline and 6 hours after ozone exposure to determine if treatment with gamma tocopherol/placebo impacts ozone-induced sputum eosinophilia.
Time Frame: baseline and 6 hours post-ozone exposure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent eosinophils
Arm/Group | Gamma Tocopherol (N=7) | Placebo (N=7)
Number analyzed (Participants) | 7 | 7
percent eosinophils | 0.8 (3.7) | -1.1 (3.0)

3. Secondary Outcome: Change in Sputum Interleukin (IL)-1b From Baseline Following Ozone Exposure
Description: Participants provide induced sputum samples before and 6 hours after Ozone exposure for measurements of inflammatory cytokines. The analysis will determine if gamma tocopherol pre-treatment reduces ozone-induced sputum inflammatory cytokine production compared to placebo pre-treatment.
Time Frame: baseline and 6 hours post ozone exposure
Population: Sufficient paired sputum supernatants from pre and post-ozone were available for analysis from 15 volunteers.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Groups:
- Gamma Tocopherol: gamma tocopherol 1400 mg, taken as two 700 mg capsules every 12 hours for a total of 4 doses
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 15 | 15
picograms per milliliter | -9.7 (65.9) | 176 (687)

4. Secondary Outcome: Change in Sputum IL-6 From Baseline Following Ozone Exposure
Description: as for outcome 3
Time Frame: baseline and 6 hours post ozone exposure
Population: Sufficient paired sputum supernatants from pre and post-ozone were available for analysis from 15 volunteers.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 15 | 15
picograms per milliliter | 58.0 (225.5) | 44.3 (128.3)

5. Secondary Outcome: Change in Sputum IL-8 From Baseline Following Ozone Exposure
Description: as for outcome 3
Time Frame: baseline and 6 hours post ozone exposure
Population: Sufficient paired sputum supernatants from pre and post-ozone were available for analysis from 12 volunteers.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 12 | 12
picograms per milliliter | -341.1 (3027) | 406.8 (2769)

6. Secondary Outcome: Change in Sputum Tumor Necrosis Factor (TNF)-Alpha From Baseline Following Ozone Exposure
Description: as for outcome 3
Time Frame: baseline and 6 hours post ozone exposure
Population: Sufficient paired sputum supernatants from pre and post-ozone were available for analysis from 13 volunteers.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 13 | 13
picograms per milliliter | -61.1 (179.1) | -301.4 (1090)

7. Secondary Outcome: Change in Sputum Mucins From Baseline Following Ozone Exposure
Description: Participants provide induced sputum samples before and 6 hours after Ozone exposure for measurements of sputum mucins to determine if gamma tocopherol pre-treatment reduces ozone-induced sputum mucins compared to placebo pre-treatment.
Time Frame: baseline and 6 hours post ozone exposure
Population: Due to improper processing of the sputum samples, analysis of mucins could not be performed.
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Whole Lung Clearance of Technetium Sulfur Colloid Particles (0-120 Minutes) From Baseline Following Ozone Exposure
Description: Whole lung clearance was measured using gamma scintigraphy and represented as mean average 120 minute clearance of inhaled technetium (99mTc) sulfur colloid particles in order to estimate the rate of airway mucociliary clearance.
Time Frame: baseline and 1 hour after exiting ozone chamber
Population: This population includes those participants who completed both arms of the study (paired assessments of MCC). One participant could not complete the whole lung clearance scan during one of the study periods and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: % clearance
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 14 | 14
% clearance | 2 (7) | 0 (7)

9. Post Hoc Outcome: Change in Central Lung Clearance of Technetium Sulfur Colloid Particles (0-30 Minutes) From Baseline Following Ozone Exposure
Description: Central lung clearance (0-30 minutes) was measured using gamma scintigraphy and represented as mean average 30 minute clearance of inhaled technetium (99mTc) sulfur colloid particles from the large bronchial airways.
Time Frame: baseline and 1 hour after exiting ozone chamber
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: % clearance
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 14 | 14
% clearance | -0.2 (8.3) | -4.3 (5.0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment until the final study visit, occurring 5-10 days after the final ozone exposure (approximately 3 months and up to 6 months). If adverse events were reported at the final study visit, the participant was followed until resolution of the event.
Description: Participants completed a standardized symptom questionnaire before ozone exposure and again at 6 and 24 hours after ozone exposure. They also completed a standardized symptom questionnaire each day while taking study treatment. Participants also had the opportunity to self-report adverse events.
Arm/Group | Gamma Tocopherol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 6/17 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gamma Tocopherol (N=17) | Placebo (N=16)
GI Distress (Gastrointestinal disorders) | 5 (6) | 1 (1) — Abdominal cramping, diarrhea, nausea,vomiting
nasal soreness (General disorders) | 1 (1) | 0 (0) — nasal turbinate soreness
URI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Upper respiratory Infection
Pain on deep inspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — pain on deep inspiration following ozone exposure
headache (General disorders) | 0 (0) | 1 (1) — headache
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Mild shortness of breath
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — self-reported wheezing on questionnaire after ozone exposure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT02911688/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT02911688/SAP_001.pdf